CLINICAL TRIAL: NCT02387177
Title: Resiliency Training for Adolescent Neurofibromatosis Patients Via Videoconferencing With Skype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Children's Tumor Foundation (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P000702
Record Dates: First submitted 2015-02-25; First posted 2015-03-12 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Neurofibromatoses
MeSH Terms: conditions — Neurofibromatoses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress Management Group 1 (Experimental): Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Interventions: Behavioral: Stress Management Group 1
- Stress Management Group 2 (Experimental): Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Interventions: Behavioral: Stress Management Group 2

INTERVENTIONS:
Behavioral: Stress Management Group 1 — Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Arms: Stress Management Group 1
Behavioral: Stress Management Group 2 — Subjects will attend group stress management sessions via Skype once weekly for 8 weeks and learn stress/NF symptoms managements techniques.
  Arms: Stress Management Group 2

SUMMARY:
The aim of this research is to adapt the NF-specific adult version of the Skype 3RP for use with adolescents, and to test its feasibility, acceptability, and preliminary effect in improving quality of life, and in decreasing stress and psychological distress.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 12 and 17
2. Can read and speak English at or above the 6th grade level
3. Diagnosis of neurofibromatosis type 1 or neurofibromatosis type 2 by a specialized medical provider

Exclusion Criteria:

1. Severe active or untreated major mental illness that would interfere with study participation, to be determined at the discretion of the study investigator (e.g. untreated psychosis or suicidality)
2. Recent (within past 3 months) change in antidepressant medication
3. Use of formal relaxation training (including past participation in a mind-body program), currently or in the past 6 months
4. Unable or unwilling to sign the informed consent documents
5. Unable or unwilling to participate in an intervention delivered via videoconferencing with Skype

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Quality of life (WHO-QOLBREFadol) | Change between Baseline (week0), Post-intervention (Week8) and Follow Up (Week 36)
  Measures quality of life

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Situations in one's life over the past month/week are appraised as stressful
The Pain Catastrophizing Scale - Child Version (PCS-C) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Measures how individuals experience pain
Patient Health Questionnaire for Adolescents (PHQ-A) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Symptoms of depression and functional impairment
Pain Interference Index (PII) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  How much pain has interfered with their life
Child and Adolescent Mindfulness Measure (CAMM) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Assesses mindfulness in children and adolescents
Interpersonal Reactivity Index (IRI) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Assesses the cognitive and affective dimensions of empathy
Epworth Sleepiness Scale-Revised for Children (ESS) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Measures how likely one is to doze off or sleep in certain situations
Gratitude Questionnaire Six-Item Form (GQ-6) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Assesses individual differences in the proneness to experience gratitude in daily life
Life Orientation Test (LOT) Optimism Scale | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Individual differences in generalized optimism versus pessimism
Functional Assessment of Chronic Illness Therapy- Spiritual Well-Being Scale (FACIT-Sp) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Spiritual well-being (sense of meaning in life and the sense of strength in one's faith) over the past 7 days
MOS (Support/Empathy) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Measures recent thinking about the various dimensions of social support.
Measure of Current Status (MOCS) Part A | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  Measures participants' current self-perceived status on several skills that are targeted by the intervention: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed.
Generalized Anxiety Disorder 7-item (GAD-7) scale | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  A brief measure for assessing generalized anxiety disorder
Quality of Life (WHOQOL-BREF) | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  The WHOQOL-BREF comprises of 26 items which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.
Satisfaction with life adolescent | Change between Baseline (week 0), Post-intervention (week 8) and Follow Up (week 32)
  measures global satisfaction with life

OTHER OUTCOMES:
Demographics | Baseline (week 0)
  Basic demographics
Expectancy Questionnaire | Baseline (week 0)
  Measures how much the participant believes the intervention will work
Intent to Attend | Baseline (week 0)
  Measures how likely and how motivated the participants is to attend the next session.
Participant Feedback - Program Satisfaction Questionnaire | Post-intervention (week 8)
  Measures how satisfied the participant is with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maira Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States